CLINICAL TRIAL: NCT01511536
Title: A Phase I/II Study of Cabazitaxel Combined With Abiraterone Acetate and Prednisone in Patients With Metastatic Castrate-Resistant Prostate Cancer (CRPC) Whose Disease Has Progressed After Docetaxel Chemotherapy
Brief Title: Cabazitaxel and Abiraterone Acetate in Patients With Metastatic Castrate-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD12128; 2011-001506-96 (EudraCT Number); U1111-1121-6324 (Other: UTN)
Record Dates: First submitted 2012-01-04; First posted 2012-01-18 (Estimated); Results first posted 2015-11-04 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1: Cabazitaxel 20 mg/m^2 + Abiraterone 1000 mg (Experimental): Cabazitaxel 20 mg/m^2 intravenous (IV) infusion on Day 1 of each 21-day cycle in combination with abiraterone acetate 1000 mg orally once daily and prednisone 5 mg orally twice daily until disease progression, unacceptable toxicity or consent withdrawal.
  Interventions: Drug: Cabazitaxel XRP6258; Drug: Abiraterone acetate; Drug: Prednisone 5 mg
- Phase 1: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg (Experimental): Cabazitaxel 25 mg/m^2 IV infusion on Day 1 of each 21-day cycle in combination with abiraterone acetate 1000 mg orally once daily and prednisone 5 mg orally twice daily until disease progression, unacceptable toxicity or consent withdrawal.
  Interventions: Drug: Cabazitaxel XRP6258; Drug: Abiraterone acetate; Drug: Prednisone 5 mg
- Phase 2: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg (Experimental): Cabazitaxel at maximum tolerated dose (MTD) as determined in phase 1 part (25 mg/m^2) IV infusion on Day 1 of each 21-day cycle in combination with abiraterone acetate 1000 mg orally once daily and prednisone 5 mg orally twice daily until disease progression, unacceptable toxicity or consent withdrawal.
  Interventions: Drug: Cabazitaxel XRP6258; Drug: Abiraterone acetate; Drug: Prednisone 5 mg

INTERVENTIONS:
Drug: Cabazitaxel XRP6258 — Pharmaceutical form:solution Route of administration: injection
Drug: Abiraterone acetate — Pharmaceutical form:tablets Route of administration: oral
Drug: Prednisone 5 mg — Route of administration: oral

SUMMARY:
Primary Objectives:

* To determine the maximum tolerated dose, and dose limiting toxicities of cabazitaxel administered as a 1-hour infusion every 3 weeks in combination with oral daily abiraterone acetate and prednisone in participants with metastatic Castrate-resistant prostate cancer (CRPC)
* To estimate the anti-tumor activity of cabazitaxel in combination with abiraterone acetate and prednisone in terms of prostate-specific antigen (PSA) response rate.

Secondary Objectives:

* To characterize the safety profile of the combination
* To evaluate the pharmacokinetic profile of cabazitaxel and abiraterone in the proposed combination and dosing schedule
* To assess preliminary antitumor activity of the combination in terms of progression-free survival, PSA progression free survival and objective response rate, and overall survival

DETAILED DESCRIPTION:
The study duration was to include a period for inclusion of up to 3 weeks and a 3-week treatment cycle(s). The participants might continue treatment until disease progression, unacceptable toxicity or willingness to stop followed by a minimum of 30-day follow-up

ELIGIBILITY:
Inclusion criteria :

* Diagnosis of prostate adenocarcinoma proven histologically or cytologically, resistant to hormone therapy and previously treated with a docetaxel-containing regimen. In Phase 2 part, participants should have been treated with abiraterone acetate for at least 3 months and should continue treatment with abiraterone acetate before study entry
* Presence of metastatic prostate cancer.
* Participant must had progressive disease documented by rising PSA defined as 2 sequential increases above a previous lowest reference value (each PSA value must be obtained at least 1 week apart. A PSA value of at least 6 ng/mL was required at study entry). In Phase 1 part, in addition to rising PSA, progressive disease must be documented by:

  1. Increase in non-measureable or measurable disease, and/or
  2. Appearance of new lesions, including those on bone scan (≥2 new lesions on 2 consecutive bone scans if progressive disease diagnosed on bone scan only) consistent with progressive prostate cancer
* Effective castration (serum testosterone levels ≤0.50 ng/mL) by orchiectomy and/or luteinizing hormone-releasing hormone agonists /antagonist.

  1. If the participant had been treated with luteinizing hormone-releasing hormone agonists/antagonist (i.e., without orchiectomy), then this therapy had been initiated at least 4 weeks prior to cycle 1 day 1 and should be continued throughout the study.
  2. Prior anti-androgen therapy should be stopped before enrollment
* Eastern Cooperative Oncology Group performance status: 0 - 1.

Exclusion criteria:

Previous treatment with mitoxantrone or cabazitaxel.

* Prior bone-seeking radio-isotope therapy (participants treated with Radium223 were not excluded from the study). Radiotherapy to ≥30% of bone marrow.
* Adverse events from any prior anticancer therapy of grade >1 at the time of enrollment.

Prior surgery, radiation, chemotherapy, or other anti-cancer therapy within 4 weeks prior to enrollment in the study (except luteinizing hormone-releasing hormone agonist /antagonist and abiraterone acetate in the Phase 2 part of the study); small field single fraction palliative radiation within 1 week.

* Prior malignancy. Curatively treated basal cell or squamous cell skin or superficial (pTis, pTa, and pT1) bladder cancer were allowed, as well as any other cancer for which chemotherapy had been completed ≥ 3 years ago and from which the participant had been disease-free for ≥ 3 years.
* Participation in another clinical trial and any concurrent treatment with any investigational drug within 30 days prior to enrollment.
* Known brain or leptomeningeal metastases.
* Any severe acute or chronic medical condition which could impair the ability of the participant to participate to the study or to comply with the study procedures or interfere with interpretation of study results.
* Other concurrent serious illness or medical conditions
* Absence of signed and dated participant informed consent form prior to enrollment into the study.
* History of hypersensitivity to docetaxel, polysorbate 80
* Known allergies, hypersensitivity or intolerance to prednisone or excipients of abiraterone acetate
* Known history of mineralocorticoid excess or deficiency
* Inadequate organ and bone marrow function
* Contraindications to the use of corticosteroid treatment.
* Symptomatic peripheral neuropathy grade > 1
* Concurrent treatment with strong inducers or strong inhibitors of cytochrome P450 (CYP450) 3A4
* Concurrent treatment with medications metabolized by cytochrome P2D6 (CYP2D6), particularly for those with a small therapeutic window
* History of cardiac arrhythmias requiring medical therapy such as atrial fibrillation requiring anticoagulation or digoxin/digitalis; uncontrolled angina pectoris. History of congestive heart failure or myocardial infarction within last 6 months was also not allowed.
* Uncontrolled hypertension (systolic BP ≥160 mmHg or diastolic BP ≥ 95 mmHg). Participants with a history of hypertension were allowed, provided that blood pressure was controlled to within these limits by anti-hypertensive treatment
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 12 months, severe or unstable angina, or New York Heart Association Class III or IV heart disease or cardiac left ventricular ejection fraction measurement of <50% at baseline
* Participants with reproductive potential who did not agree to use accepted and effective method of contraception in conjunction with their partner(s) during the study treatment period.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-03; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- United States (2):
  - Investigational Site Number 840001, San Francisco, California
  - Investigational Site Number 840002, New Haven, Connecticut
- Investigational Site Number 250001, Villejuif, France
- Investigational Site Number 826001, Sutton, United Kingdom

REFERENCES:
- [Derived] Massard C, Mateo J, Loriot Y, Pezaro C, Albiges L, Mehra N, Varga A, Bianchini D, Ryan CJ, Petrylak DP, Attard G, Shen L, Fizazi K, de Bono J. Phase I/II trial of cabazitaxel plus abiraterone in patients with metastatic castration-resistant prostate cancer (mCRPC) progressing after docetaxel and abiraterone. Ann Oncol. 2017 Jan 1;28(1):90-95. doi: 10.1093/annonc/mdw441. PMID 28039155
- [Derived] Huang X, Chau CH, Figg WD. Challenges to improved therapeutics for metastatic castrate resistant prostate cancer: from recent successes and failures. J Hematol Oncol. 2012 Jul 2;5:35. doi: 10.1186/1756-8722-5-35. PMID 22747660

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 2 centers in phase 1 part and 3 centers in phase 2 part between March 2012 and April 2014.
Pre-assignment Details: Phase I was a dose escalation part of Cabazitaxel, administered with a constant dose of abiraterone, to determine maximally tolerated dose. Phase 2 was efficacy and safety evaluation of Cabazitaxel at a dose, determined in Phase 1, in combination with abiraterone.
Period: Phase 1
Arm/Group | Phase 1: Cabazitaxel 20 mg/m^2 + Abiraterone 1000 mg | Phase 1: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg | Phase 2: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg
Started | 3 | 7 | 0 (Phase 1 and phase 2 are separate populations.)
Completed | 3 (Cancer progression,adverse event,consent withdrawal are considered as completed(defined in protocol)) | 6 (Cancer progression,adverse event,consent withdrawal are considered as completed(defined in protocol)) | 0
Not Completed | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0
Period: Phase 2
Arm/Group | Phase 1: Cabazitaxel 20 mg/m^2 + Abiraterone 1000 mg | Phase 1: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg | Phase 2: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg
Started | 0 | 0 | 27
Completed | 0 | 0 | 18 (Cancer progression,adverse event,consent withdrawal are considered as completed(defined in protocol))
Not Completed | 0 | 0 | 9
Not completed — Other | 0 | 0 | 9

BASELINE CHARACTERISTICS:
Population: All treated/safety population defined as all registered participants exposed to both investigational medicinal product (IMP) components, regardless of the amount of treatment administered.
Groups:
- Phase 1: Cabazitaxel 20 mg/m^2 + Abiraterone 1000 mg: Cabazitaxel 20 mg/m^2 IV infusion on Day 1 of each 21-day cycle in combination with abiraterone acetate 1000 mg orally once daily and prednisone 5 mg orally twice daily until disease progression, unacceptable toxicity or consent withdrawal.
- Phase 2: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg: Cabazitaxel at MTD as determined in phase 1 part (25 mg/m^2) IV infusion on Day 1 of each 21-day cycle in combination with abiraterone acetate 1000 mg orally once daily and prednisone 5 mg orally twice daily until disease progression, unacceptable toxicity or consent withdrawal.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Cabazitaxel 20 mg/m^2 + Abiraterone 1000 mg | Phase 1: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg | Phase 2: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg | Total
Number analyzed (Participants) | 3 | 7 | 27 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (7.0) | 60.0 (10.0) | 67.1 (5.4) | 66.1 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 3 | 7 | 27 | 37

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximally Tolerated Dose (MTD) of Cabazitaxel in Combination With Abiraterone Acetate
Description: MTD was defined as highest dose level of cabazitaxel in combination with abiraterone acetate at which no more than 1 participant experienced dose limiting toxicities (DLT). DLT was defined as any of the following events related to study treatment: 1) Grade 3 or 4 non-hematological related adverse event with exception of Grade 3 fever without documented infection; Grade 3 nausea, vomiting, or diarrhea in the absence of effective maximal therapy; and Grade 3 hypersensitivity reaction in the absence of required premedication. 2) Hematological toxicity: Febrile neutropenia (fever of unknown origin ≥38.5°C with neutropenia Grade 3 or 4); Neutropenia Grade 4 lasting >7 days; Thrombocytopenia Grade 4 or Grade 3 complicated by hemorrhage. 3) Re-treatment delay of more than 2 weeks due to delayed recovery from a toxicity related to study treatment to baseline or ≤ Grade 1 (except for alopecia). Grades were based on National Cancer Institute CommonTerminology Criteria for Adverse Events v4.03.
Time Frame: Up to Cycle 2 of Phase 1 (up to 42 days)
Population: Analysis was performed on DLT evaluable population defined as all participants who received the first 2 cycles, unless they discontinued the study drug during the first 2 cycles for a DLT.
Measure: Number; unit: mg/m^2
Groups:
- Phase 1: Overall Population: Cabazitaxel 20 or 25 mg/m^2 IV infusion on Day 1 of each 21-day cycle in combination with abiraterone acetate 1000 mg orally once daily and prednisone 5 mg orally twice daily until disease progression, unacceptable toxicity or consent withdrawal.
Arm/Group | Phase 1: Overall Population
Number analyzed (Participants) | 9
mg/m^2 | 25

2. Primary Outcome: Phase 2: Percentage of Participants With Prostate Specific Antigen (PSA) Response
Description: Prostate specific antigen (PSA) response was defined as ≥50% decrease from baseline in serum PSA levels, confirmed at least 3 weeks later. Increases of any magnitude during the first 12 weeks were ignored in determining PSA response. PSA was to be measured at baseline, every 3 weeks, throughout study period, until progression. PSA progression was defined as: -An increase of 25% above the nadir (at least 2 ng/mL), confirmed by a second PSA value at least 3 weeks apart, in participants who have achieved a ≥50% decline of PSA. -An increase in PSA by 25 % above the baseline level (at least 2 ng/mL), confirmed by a second PSA value at least 3 weeks apart, in participants who have not achieved a ≥50% decline of PSA.
Time Frame: Baseline, every 3 weeks up to PSA progression (maximum duration: 603 days)
Population: Analysis was performed on efficacy/activity population included all participants who had received at least 2 cycles of the study drug in Phase 2, and had a baseline and at least one post-baseline assessment for the efficacy variable of interest.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg
Number analyzed (Participants) | 26
percentage of participants | 46.2 [26.6 to 66.6]

3. Secondary Outcome: Phase 2: Objective Progression Free Survival (PFS)
Description: Objective PFS was defined as the time interval between the date of enrollment and the first occurrence of any of the events:
  1) Radiological tumor progression (assessed using Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1) was defined as at least a 20 percent increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions and/or unequivocal progression of existing non target-lesions. in case of progressive disease (PD) diagnosed only on non target bone lesions on bone scan, PD was to be considered only in case of appearance of at least 2 new lesions on bone scan confirmed 6 weeks later by another bone scan, and at least the appearance of 2 new additional lesions. 2) Death due to any cause.
  Analysis was performed by Kaplan-Meier method.
Time Frame: From baseline until radiological tumor or disease progression or death due to any cause, assessed up to Month 5
Population: Analysis was performed on efficacy/activity population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg
Number analyzed (Participants) | 26
months | NA [4.731 to NA] — Data was not calculable as <50% participants had event of interest.

4. Secondary Outcome: Phase 2: PSA Progression Free Survival
Description: Prostate-specific antigen progression-free survival was defined as the time interval between the date of treatment start and the date of either first documented PSA progression or death due to any cause, whichever was earlier. PSA was to be measured at baseline, every 3 weeks, throughout study period, until progression. PSA progression was defined as: -An increase of 25% above the nadir (at least 2 ng/mL), confirmed by a second PSA value at least 3 weeks apart, in participants who have achieved a ≥50% decline of PSA. -An increase in PSA by 25 % above the baseline level (at least 2 ng/mL), confirmed by a second PSA value at least 3 weeks apart, in participants who have not achieved a ≥50% decline of PSA.
  Analysis was performed by Kaplan Meire method.
Time Frame: Baseline, every 3 weeks up to PSA progression (maximum duration: 603 days)
Population: Analysis was performed on efficacy/activity population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg
Number analyzed (Participants) | 26
months | 6.93 [4.140 to 10.251]

5. Secondary Outcome: Phase 2: Percentage of Participants With Objective Response
Description: Objective response was defined as having complete response (CR) or Partial Response (PR) assessed by RECIST 1.1. CR was defined as disappearance of all target, non-target lesions; normalization of tumor marker level and all lymph nodes size was <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters).
Time Frame: Baseline, every 12 weeks there after until disease progression (maximum duration: 603 days)
Population: Efficacy/activity population. Number of participants analyzed=participants with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg
Number analyzed (Participants) | 14
percentage of participants | 21.4 [4.7 to 50.8]

6. Secondary Outcome: Phase 2: Overall Survival
Description: Overall survival was defined as the time interval from the date of treatment start to the date of death due to any cause. In absence of confirmation of death, survival time was censored at the earlier of the last date the participant was known to be alive and the study cut-off date. Analysis was performed by Kaplan-Meier method.
Time Frame: From baseline up to death or study cut-off (maximum duration: 603 days)
Population: Analysis was performed on efficacy/activity population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg
Number analyzed (Participants) | 26
months | NA [9.429 to NA] — Data was not calculable as <50% participants had event of interest.

7. Secondary Outcome: Phase 2: Pharmacokinetic of Cabazitaxel : Maximum Plasma Concentration Observed (Cmax)
Time Frame: 5 minutes before cabazitaxel infusion; at end of cabazitaxel infusion; 0.25 hours post-cabazitaxel infusion; any time between 1 to 4 hours, between 6 to 24 hours, between 48 to 96 hours post cabazitaxel infusion on Day 1-Cycle 1
Population: Analysis was performed on pharmacokinetic (PK) population which included all participants who received at least 1 treatment. Pre-dose samples from 3 participants of Phase 2, were above lower limit of quantification (LLOQ) (1.00 ng/mL). Hence, those participants were excluded from analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 2: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg
Number analyzed (Participants) | 24
ng/mL | 330 (187)

8. Secondary Outcome: Phase 2: Pharmacokinetic of Cabazitaxel : Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: Area under the concentration-time curve calculated using the following equation: AUC = Plasma clearance (CL)/dose
Time Frame: as for outcome 7
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Phase 2: Cabazitaxel 25 mg/ m^2 + Abiraterone 1000 mg: Cabazitaxel at MTD as determined in phase 1 part (25 mg/m^2) IV infusion on Day 1 of each 21-day cycle in combination with abiraterone acetate 1000 mg orally once daily and prednisone 5 mg orally twice daily until disease progression, unacceptable toxicity or consent withdrawal.
Arm/Group | Phase 2: Cabazitaxel 25 mg/ m^2 + Abiraterone 1000 mg
Number analyzed (Participants) | 24
ng*h/mL | 817 (117)

9. Secondary Outcome: Phase 2: Pharmacokinetic of Cabazitaxel : Terminal Half-life (t 1/2z)
Time Frame: as for outcome 7
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Phase 2: Cabazitaxel 25 mg/ m^2 + Abiraterone 1000 mg
Number analyzed (Participants) | 24
hour | 91.6 (62.6)

10. Secondary Outcome: Phase 2: Pharmacokinetic of Cabazitaxel : Total Plasma Clearance (CL)
Time Frame: as for outcome 7
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: L/h/m^2
Arm/Group | Phase 2: Cabazitaxel 25 mg/ m^2 + Abiraterone 1000 mg
Number analyzed (Participants) | 24
L/h/m^2 | 31.4 (4.67)

11. Secondary Outcome: Phase 2: Pharmacokinetic of Cabazitaxel : Volume of Distribution at Steady State (Vss)
Time Frame: as for outcome 7
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: L/m^2
Arm/Group | Phase 2: Cabazitaxel 25 mg/ m^2 + Abiraterone 1000 mg
Number analyzed (Participants) | 24
L/m^2 | 2711 (2493)

12. Secondary Outcome: Phase 2: Pharmacokinetic of Abiraterone : Maximum Plasma Concentration Observed (Cmax)
Time Frame: 0 hour (before abiraterone administration); 1, 2, 4, 6, 8, 12, 24 hours post abiraterone administration on Day 1-Cycle 1
Population: Analysis was performed on PK population. One participant was excluded from analysis due to aberrant data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 2: Cabazitaxel 25 mg/ m^2 + Abiraterone 1000 mg
Number analyzed (Participants) | 26
ng/mL | 216 (152)

13. Secondary Outcome: Phase 2: Pharmacokinetic of Abiraterone : First Time to Reach Cmax (Tmax)
Time Frame: as for outcome 12
Population: Analysis was performed on PK population. One participant was excluded from analysis due to aberrant data.
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 2: Cabazitaxel 25 mg/ m^2 + Abiraterone 1000 mg
Number analyzed (Participants) | 26
hour | 2.00 [1.00 to 6.00]

14. Secondary Outcome: Phase 2: Pharmacokinetic of Abiraterone : Area Under the Plasma Concentration Versus Time Curve From Time 0 to 24 Hours (AUC 0-24)
Description: Area under the plasma concentration-time curve calculated using the trapezoidal method from time zero to 24 hours corresponding to abiraterone acetate dosing interval.
Time Frame: as for outcome 12
Population: Analysis was performed on PK population. One participant was excluded from analysis due to aberrant data.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Phase 2: Cabazitaxel 25 mg/ m^2 + Abiraterone 1000 mg
Number analyzed (Participants) | 26
ng*h/mL | 928 (466)

15. Secondary Outcome: Phase 2: Pharmacokinetic of Abiraterone : Concentration Observed Just Before Treatment Administration During Repeated Dosing at Steady State (Ctrough ss)
Time Frame: Pre abiraterone dose on Day 1 of Cycle 1
Population: Analysis was performed on PK population. One participant was excluded from analysis due to aberrant data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 2: Cabazitaxel 25 mg/ m^2 + Abiraterone 1000 mg
Number analyzed (Participants) | 26
ng/mL | 9.99 (13.0)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (603 days) regardless of seriousness or relationship to investigational product
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during 'on treatment period' (time from first dose of study drug [cabazitaxel or abiraterone, whichever came first] to last dose of study drug [cabazitaxel or abiraterone, whichever came last] + 30 days). Analysis was performed on safety population.
Arm/Group | Phase 1: Cabazitaxel 20 mg/m^2 + Abiraterone 1000 mg | Phase 1: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg | Phase 2: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg
Serious Adverse Events (participants affected / at risk) | 3/3 | 4/7 | 21/27
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Cabazitaxel 20 mg/m^2 + Abiraterone 1000 mg (N=3) | Phase 1: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg (N=7) | Phase 2: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg (N=27)
Device related infection (Infections and infestations) | 0 | 0 | 1
Neutropenic infection (Infections and infestations) | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1
Parasitic gastroenteritis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 3
Spinal cord infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 4
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Anuria (Renal and urinary disorders) | 0 | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 3
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 4
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 3
Urinary retention (Renal and urinary disorders) | 0 | 0 | 2
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 2
Disease progression (General disorders) | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Cabazitaxel 20 mg/m^2 + Abiraterone 1000 mg (N=3) | Phase 1: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg (N=7) | Phase 2: Cabazitaxel 25 mg/m^2 + Abiraterone 1000 mg (N=27)
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2
Oral candidiasis (Infections and infestations) | 0 | 1 | 1
Oral fungal infection (Infections and infestations) | 0 | 1 | 2
Tinea pedis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 3
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 13
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 7
Affective disorder (Psychiatric disorders) | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 4
Headache (Nervous system disorders) | 1 | 0 | 3
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 2 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 2
Syncope (Nervous system disorders) | 0 | 1 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 2 | 2
Hot flush (Vascular disorders) | 1 | 2 | 1
Hypotension (Vascular disorders) | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 15
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1
Gastrointestinal hypermotility (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 4
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 5 | 14
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 5
Toothache (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 5
Hair disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 2 | 8
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Asthenia (General disorders) | 2 | 3 | 16
Fatigue (General disorders) | 0 | 1 | 2
Granuloma (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 4
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 3
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 13
Weight increased (Investigations) | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.